CLINICAL TRIAL: NCT07188389
Title: Immunometabolism of Exercise and Fitness
Brief Title: Immunometabolism of Exercise
Acronym: IMEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Emily C Lavoy, Associate Professor, University of Houston
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00004272
Record Dates: First submitted 2025-09-17; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Cardiorespiratory Fitness and Acute Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acute effects: Moderate Intensity Exercise (Experimental): Participants with a moderate fitness level (determined by VO2max value recorded during graded exercise test) will cycle 30minutes exercise below ventilatory threshold. Outcome measures will be compared within-subject across blood sampled before exercise, immediately after exercise, and 2h post exercise. The order of the exercise sessions (above vs below threshold) will be randomized.
  Interventions: Behavioral: Acute exercise-moderate intensity
- Acute effects: Heavy intensity exercise (Experimental): Participants with a moderate fitness level (determined by VO2max value recorded during graded exercise test) will bicycle 30 minutes above ventilatory threshold. Outcome measures will be compared within-subject across blood sampled before exercise, immediately after exercise, and 2h post exercise. The order of the exercise sessions (above vs below threshold) will be randomized.
  Interventions: Behavioral: Acute effects-heavy intensity

INTERVENTIONS:
Behavioral: Acute exercise-moderate intensity — 30 minutes of cycling exercise at moderate (90% of first ventilatory threshold)
  Arms: Acute effects: Moderate Intensity Exercise
Behavioral: Acute effects-heavy intensity — Participants will cycle 30 minutes at heavy (110% of first ventilatory threshold) intensity
  Arms: Acute effects: Heavy intensity exercise

SUMMARY:
This study aims to examine the effects of acute aerobic exercise and cardiorespiratory fitness on cellular metabolism of CD8+ T cells and regulatory T cells (Tregs) found in the peripheral blood of humans. In addition, the study will investigate whether the effects of exercise differ based on exercise intensity, as well as whether the effects of exercise and fitness differ between subpopulations of CD8+ T cells and Tregs. Finally, the study aims to examine whether exercise- and fitness-induced changes in cell metabolism relate to changes in cell function.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 20-40 years
* individuals presenting with average (40th-60th percentile) cardiorespiratory fitness (i.e., VO2max/VO2peak) for their age and sex will be included in acute exercise experiments; individuals with VO2max/VO2peak value >20ml/kg/min will be included in cardiorespiratory fitness experiments
* individuals categorized as 'low risk' for a cardiovascular event/heart disease when screened by American College of Sports Medicine (ACSM) criteria

Exclusion Criteria:

* adults under the age of 20 and over the age of 40
* Individuals with contraindications to exercise testing will be excluded
* Individuals with musculoskeletal impairments preventing them from exercising on a cycle ergometer
* Individuals with disease history known to impact the immune system and/or systemic metabolism will be excluded, including autoimmune diseases, HIV, Hepatitis, diabetes, cancer (completed treatment within <6 months prior), hyper- or hypothyroidism
* Pregnancy
* Individuals using medications known to impact the cardiopulmonary and/or immune response to exercise with be excluded, including those using medication to control blood pressure (e.g., beta-blockers), daily steroidal and nonsteroidal anti-inflammatories (except daily aspirin), prescription allergy medication, ADHD medication (Ritalin or Adderall), thyroid medication (e.g., Levothyroxine), and chemotherapy (including treatments within the last 6 months).
* Individuals habitually using tobacco products within the last 6 months or with excessive alcohol intake (>10 drinks/week)

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Metabolic Function | At rest, immediately after, and two hours after exercise
  Cellular metabolic activity and poise of T cells as measured by flow cytometry (SCENITH)
Immune Cell function | At rest, immediately after, and two hours after exercise
  Stimulated IFN-gamma, perforin and IL-10 production, as measured by flow cytometry
Metabolic Regulation | At rest, immediately after, and two hours after exercise
  Expression of genes involved in cellular energy metabolism, as assessed by RT-PCR
Mitochondrial Regulation | At rest, immediately after, and two hours after exercise
  Mitochondrial mass and membrane potential, as assessed by flow cytometry

SECONDARY OUTCOMES:
Peripheral immune cell composition | At rest, immediately after, and two hours after exercise
  Number (concentration) of immune cell subsets in peripheral blood, as measured by hematology analyzer and flow cytometer

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided